CLINICAL TRIAL: NCT03032302
Title: Micronutrient Intervention Effects on Cognitive Outcomes in Post-Acute Traumatic Brain Injury
Brief Title: Micronutrient Supplement Effects on Cognitive Outcomes in Post-Acute TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Collaborators: Sheffield Teaching Hospitals NHS Foundation Trust (Other); Rotherham Doncaster and South Humber NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: STH19529
Record Dates: First submitted 2016-12-22; First posted 2017-01-26 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Traumatic Brain Injury
Keywords: TBI
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multivitamin (Experimental): Swisse Womens 50+ Ultivite Multivitamin. Once daily.
  Interventions: Dietary Supplement: Swisse Womens 50+ Ultivite Multivitamin; Dietary Supplement: Holland and Barrett Triple Strength Omega-3 Fish Oil
- Omega-3 Fatty Acids (Experimental): Holland and Barrett Triple Strength Omega-3 Fish Oils. Once Daily
  Interventions: Dietary Supplement: Swisse Womens 50+ Ultivite Multivitamin; Dietary Supplement: Holland and Barrett Triple Strength Omega-3 Fish Oil
- Control (No Intervention): Treatment as usual (cognitive rehabilitation, occupational therapy, physiotherapy; as required)

INTERVENTIONS:
Dietary Supplement: Swisse Womens 50+ Ultivite Multivitamin — Single tablet taken once daily
  Arms: Multivitamin; Omega-3 Fatty Acids
Dietary Supplement: Holland and Barrett Triple Strength Omega-3 Fish Oil — Single capsule taken once daily
  Arms: Multivitamin; Omega-3 Fatty Acids

SUMMARY:
Traumatic brain injury (TBI) refers to neuronal damage occurring as the result of an external force being applied to brain tissue. In the United Kingdom annual figures (2013-2014) show 449,000 hospital admittances with a diagnosis of head injury with males up to five times more likely to sustain a head injury than females. Traumatic brain injury (TBI) causes life-long disability, with no significant reduction in life expectancy, affecting a diverse range of cognitive and social functions including memory, task planning and execution, impulse control, social interactions, personality changes and depression. Following traumatic brain injury acquired deficits can lead to problems with resumption of aspects of daily life, particularly in terms of returning to work and interpersonal relationships.

The initial injury triggers a secondary cascade of metabolic, neurochemical and cellular changes within the brain, primarily aimed at limiting damage and stimulating repair. Paradoxically prolonged secondary cascade mechanisms, including haemorrhage, oedema, neuroinflammation and axonal injury, results in exacerbation of deficits observed. The heterogeneous on-going nature of the secondary cascade presents clinicians with opportunities to intervene in an attempt to limit neuronal damage. A large body of nutritional research has been focused on addressing the hypermetabolic and catabolic states created by secondary cascade processes in the acute stage. Addressing these demands has played a significant role in reducing mortality and infection rates following head injury, however there has not been the same depth of research investigating the post-acute period (once individuals are discharged from hospital).

DETAILED DESCRIPTION:
Micronutrients (including vitamins, minerals and certain polyunsaturated fatty acids) are required by the brain for normal functioning and, with few exceptions, can only be obtained through dietary sources. Research into degenerative diseases of aging have linked mitochondrial aging and DNA damage caused by micronutrient deficiency to greater incidence of cognitive decline and stroke, among other diseases, in the general population, particularly in those consuming food rich in fats and carbohydrates but poor in micronutrient content. Other research focusing on cognition, behaviour and mood state has associated micronutrient deficiencies with a wide range of neurological conditions including Alzheimer's Disease, Parkinson's Disease, multiple sclerosis, autism spectrum disorders, depression, fatigue and schizophrenia. There have however been very few studies using micronutrient interventions in post-acute human TBI. In a study with thirty retired American Football players an intervention including supplementation with a broad-spectrum multivitamin, omega-3 fish oils and a number of other substances resulted in significant percentile score improvements in almost half of the participants (n=100) across a broad range of cognitive measures. Findings demonstrated that micronutrient intervention can result in significant measurable improvements in those with TBI many years following the initial insult. A normative study will be conducted with three groups assigned to Vit D, Vit C and multivitamin arms (N = 60) tested at baseline on cognitive function and post-intervention. The TBI study will recruit three groups of individuals with post-acute traumatic brain injuries and measure whether there is improved cognitive outcomes (measured by test-retest on a cognitive battery) associated with the supplements shown to be most effective in the pilot study.

ELIGIBILITY:
Inclusion Criteria:

* First and only traumatic brain injury.
* Complex mild to moderate injury.
* 3-24 months post-injury

Exclusion Criteria:

* Unable to give informed consent.
* Already taking micronutrient/fatty acid supplements.
* Hemianopia
* Hemiplegia.
* Pregnant or breastfeeding.
* Diagnosed with clinically low blood pressure, diabetes, or disease of neurodegeneration.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-04-18 (Actual); Study Completion 2020-04-18 (Actual)

PRIMARY OUTCOMES:
Performance on cognitive test measures (a battery of standardized tests; memory, executive function, social cognition, general intelligence, learning and processing speed) | Three time points: baseline (T1), 8 weeks (T2) and 22 weeks (T3)
  Analysis of change in cognitive test battery results between each time point (T2 minus T1. T3 minus T2. T3 minus T1)

SECONDARY OUTCOMES:
Average dietary intake of micronutrients and fatty acids | Data collected at four time points (3 day diaries) during participant's involvement in the study via participants filling in paper food diary
  Analysis of dietary intake via Nutritics software (https://www.nutritics.com/p/references), average intake value for each micronutrient supplied by software output. This will be compared to recommended daily amounts to evaluate levels of sufficiency/insufficiency in each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Lynne A Barker, PhD, Study Director — Sheffield Hallam University
Locations (1):
- Sheffield Hallam University, Sheffield, South Yorkshire, United Kingdom

REFERENCES:
- [Background] Lippert-Gruner M, Kuchta J, Hellmich M, Klug N. Neurobehavioural deficits after severe traumatic brain injury (TBI). Brain Inj. 2006 Jun;20(6):569-74. doi: 10.1080/02699050600664467. PMID 16754282
- [Background] Bombardier CH, Fann JR, Temkin NR, Esselman PC, Barber J, Dikmen SS. Rates of major depressive disorder and clinical outcomes following traumatic brain injury. JAMA. 2010 May 19;303(19):1938-45. doi: 10.1001/jama.2010.599. PMID 20483970
- [Background] Borzotta AP, Pennings J, Papasadero B, Paxton J, Mardesic S, Borzotta R, Parrott A, Bledsoe F. Enteral versus parenteral nutrition after severe closed head injury. J Trauma. 1994 Sep;37(3):459-68. doi: 10.1097/00005373-199409000-00022. PMID 8083910
- [Background] Cook AM, Peppard A, Magnuson B. Nutrition considerations in traumatic brain injury. Nutr Clin Pract. 2008 Dec-2009 Jan;23(6):608-20. doi: 10.1177/0884533608326060. PMID 19033220
- [Background] Ames BN. Optimal micronutrients delay mitochondrial decay and age-associated diseases. Mech Ageing Dev. 2010 Jul-Aug;131(7-8):473-9. doi: 10.1016/j.mad.2010.04.005. Epub 2010 Apr 24. PMID 20420847
- [Background] Balion C, Griffith LE, Strifler L, Henderson M, Patterson C, Heckman G, Llewellyn DJ, Raina P. Vitamin D, cognition, and dementia: a systematic review and meta-analysis. Neurology. 2012 Sep 25;79(13):1397-405. doi: 10.1212/WNL.0b013e31826c197f. PMID 23008220
- [Background] Bitarafan S, Harirchian MH, Nafissi S, Sahraian MA, Togha M, Siassi F, Saedisomeolia A, Alipour E, Mohammadpour N, Chamary M, Honarvar NM, Saboor-Yaraghi AA. Dietary intake of nutrients and its correlation with fatigue in multiple sclerosis patients. Iran J Neurol. 2014;13(1):28-32. PMID 24800044
- [Background] Nimitphong H, Holick MF. Vitamin D, neurocognitive functioning and immunocompetence. Curr Opin Clin Nutr Metab Care. 2011 Jan;14(1):7-14. doi: 10.1097/MCO.0b013e3283414c38. PMID 21102318
- [Background] Oudshoorn C, Mattace-Raso FU, van der Velde N, Colin EM, van der Cammen TJ. Higher serum vitamin D3 levels are associated with better cognitive test performance in patients with Alzheimer's disease. Dement Geriatr Cogn Disord. 2008;25(6):539-43. doi: 10.1159/000134382. Epub 2008 May 26. PMID 18503256
- [Background] Amen DG, Wu JC, Taylor D, Willeumier K. Reversing brain damage in former NFL players: implications for traumatic brain injury and substance abuse rehabilitation. J Psychoactive Drugs. 2011 Jan-Mar;43(1):1-5. doi: 10.1080/02791072.2011.566489. PMID 21615001
- [Derived] Lucke-Wold B, Zasler ND, Ruchika F, Weisman S, Le D, Brunicardi J, Kong I, Ghumman H, Persad S, Mahan D, Delawan M, Shah S, Aghili-Mehrizi S. Supplement and nutraceutical therapy in traumatic brain injury. Nutr Neurosci. 2025 Jun;28(6):709-743. doi: 10.1080/1028415X.2024.2404782. Epub 2024 Dec 30. PMID 40440029
- See also: Nutritics — https://www.nutritics.com/p/references